CLINICAL TRIAL: NCT02698553
Title: An Open-label, Fixed Sequence Study to Evaluate Pharmacokinetics, Safety and Tolerability of Single and Repeated Dose of Extended-release Bupropion Hydrochloride (Bupropion XL) Tablets 150 mg and 300 mg Once Daily in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate Pharmacokinetics, Safety and Tolerability of Extended-release Bupropion Hydrochloride Tablets in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114883
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Depressive Disorder, Major
Keywords: Major depressive disorder; Extended release Bupropion
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion XL once daily (Experimental): Healthy subjects will receive Bupropion XL 150milligram (mg) once daily for 5 days (Day 1 to Day 5) and then Bupropion XL 300 mg once daily from Day 6 to Day 14.
  Interventions: Drug: Bupropion HCl XL tablet 150mg; Drug: Bupropion HCl XL tablet 300mg

INTERVENTIONS:
Drug: Bupropion HCl XL tablet 150mg — The 150 mg of tablet will be given to subject once daily orally. Subject will be instructed to swallow whole tablet with 240 ml of water, without crushed, divided or chewed.
Drug: Bupropion HCl XL tablet 300mg — The 300 mg of tablet will be given to subject once daily orally. Subject will be instructed to swallow whole tablet with 240 ml of water, without crushed, divided or chewed.

SUMMARY:
Bupropion is used in psychological disorder mainly in major depressive disorder (MDD). In China, buproprion Immediate Release (IR) and Sustained Release (SR) tablet have been in market for the treatment of MDD. Bupropion Hydrochloride (HCl) Extended Release (XL) tablets formulation is proposed for marketing approval in China for same indication. Therefore, a pharmacokinetic study is planned to be conducted in Chinese subjects. It is an open label, single-centre and single cycle study to evaluate the pharmacokinetics, safety and tolerability of 150 milligram (mg) and 300 mg following single and repeated daily doses. Approximately 16 males and females Chinese healthy subjects will be enrolled into the study to get 12 completed subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to actively communicate with the investigator and to complete the study-related documents; able to understand the contents of the Informed consent form (ICF) and to sign a written ICF prior to any study-specific procedures.
* Males and females aged between 18 and 45 years inclusive, at the time of signing the informed consent.
* Non-smoking healthy males and females as assessed by medical history and physical examination. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters which are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight>=50 kilograms (Kg) and Body mass index (BMI) 19.0 to 25.0 kg/square meter (m^2).
* A female subject is eligible to participate if she is of: Child-bearing potential with negative pregnancy test as determined by serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing and agrees to use the contraception methods during the study and until follow up contact.
* Male subjects with female partners of child-bearing potential must agree to use the contraception methods during the study and until follow up contact.
* ALT, ALP and total bilirubin =<1.5x upper limit of normal (ULN) (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Based on single or averaged corrected QT interval (QTc) values of triplicate ECGs obtained over a brief recording period: QTc <450 milliseconds (msec) or QTc <480 msec in subjects with bundle branch block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Drug or alcohol abuse or dependency within one year prior to enrolment. History of regular alcohol consumption within 6 months of the study, defined as: an average weekly intake of >14 drinks. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 millilitre [ml]) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Unstable disease conditions; any laboratory measurements assessed by the investigator as clinically relevant (including electroencephalogram [EEG], ECG, haematology, biochemistry and urine analysis, etc.); any disorder that might interfere with the absorption, distribution, metabolism or excretion of the study drug; or in the investigator's opinion the disease may lead to safety concerns or interfere with the pharmacokinetics assessment.
* Subjects with concurrent or previous neuropsychological disorders, as assessed by Columbia Suicidality Severity Rating (CSSR) Scale or by the investigator, have suicidal tendency, or have committed suicidal behavior/attempt.
* Known history of cerebral trauma, previous cerebral disorders, seizures or eating disorder, and other conditions that in the investigator's opinion may increase the risk of seizures.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Other Criteria
* Serum human immunodeficiency virus (HIV) antibody or Syphilis antibody positive.
* A positive pre-study drug/alcohol screen.
* Blood donation in the 3 months prior to enrolment. Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Obvious evidence of active haematological diseases, or significant blood loss in the last 3 months. History of sensitivity to heparin or heparin-induced thrombocytopenia.
* The subject has participated in a clinical trial and has received an investigational product within 30 days prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Known allergy to Bupropion Extended-Release Tablets or any of its components.
* Lactating females or women of child bearing potential used oral or implanted contraceptives within the 30 days prior to enrolment, or received injections of chronically acting contraceptives in the 1 year prior to study initiation.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Other conditions which, in the Investigator's judgment, render subjects unsuitable for the clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Time taken to reach peak plasma concentration (Tmax) of Bupropion HCl and its metabolites after single dose. | Day 1 and Day 2.
  Blood sample will be collected at pre-dosing, and 2, 3, 4, 5, 6, 8, 12, 16, and 24 hour (h) post dose.
Maximum observed concentration (Cmax) in plasma of Bupropion HCl and its metabolites after single dose. | Day 1 and Day 2.
  Blood sample will be collected at pre-dosing, and 2, 3, 4, 5, 6, 8, 12, 16, and 24 h post dose.
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC [0-24]) of Bupropion HCl and its metabolites after single dose. | Day 1 and Day 2.
  Blood sample will be collected at pre-dosing, and 2, 3, 4, 5, 6, 8, 12, 16, and 24 h post dose.
Tmax in plasma of Bupropion HCl and its metabolites after repeated doses | Day 5 to Day 19 .
  Blood sample will be collected at pre-dosing, and 2, 5, 8 and 12h post dose after 150 mg dose (Day 5) and first 300 mg (Day 6) dose respectively. Blood sample will be also collected at pre-dosing, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 h post dose after 300 mg dose (Day 14 to 19).
Steady state concentration (Css)-Css Minimum (Css_min), Css Maximum (Css_max), Average Css (Css_av) in plasma of Bupropion HCl and its metabolites after repeated dose. | Day 5 to Day 19.
  Blood sample will be collected at pre-dosing, and 2, 5, 8 and 12h post dose after 150 mg dose (Day 5) and first 300 mg (Day 6) dose respectively, and pre-dosing, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 h post dose after last 300 mg dose (Day 14 to 19).
Elimination half-life (t ½) in plasma of Bupropion HCl and its metabolites after repeated dose. | Day 5 to Day 19.
  Blood sample will be collected at pre-dosing, and 2, 5, 8 and 12 h post dose after 150 mg dose (Day 5) and first 300 mg (Day 6) dose respectively, and pre-dosing, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 h post dose after last 300 mg dose (Day 14 to 19).
Apparent clearance (CL/F) in plasma of Bupropion HCl and its metabolites after repeated dose. | Day 5 to Day 19.
  Blood sample will be collected at pre-dosing, and 2, 5, 8 and 12 h post dose after last 150 mg dose (Day 5) and first 300 mg (Day 6) dose respectively, and pre-dosing, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 h post dose after last 300 mg dose (Day 14 to 19).
Area under the concentration-time curve over the dosing interval (AUC [0-tau]) in plasma of Bupropion HCl and its metabolites after repeated dose. | Day 5 to Day 19.
  Blood sample will be collected at pre-dosing, and 2, 5, 8 and 12 h post dose after 150 mg dose (Day 5) and first 300 mg (Day 6) dose respectively, and pre-dosing, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 h post dose after last 300 mg dose (Day 14 to 19).

SECONDARY OUTCOMES:
Number of subjects with adverse event (AE) and serious adverse event (SAE). | Up to Day 33.
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Number of subjects with abnormal Haematology parameters as a measure of safety. | Up to Day 19.
  Blood sample will be collected at screening, Day 1, Day 6 and Day 19 to assess platelet counts, red blood cells (RBC) count, haemoglobin, hematocrit, white blood cells (WBC) count, reticulocyte count, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), composite of WBC differential counts.
Number of subjects with abnormal Clinical chemistry parameters as a measure of safety. | Up to Day 19.
  Blood sample will be collected at screening, Day 1, Day 6 and Day 19 to analyze blood urea nitrogen (BUN), creatinine, lactate dehydrogenase (LDH), urea, glucose level (fasting), composite electrolytes levels, gamma-glutamyl transferase (GGT), aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase (ALP) levels, total cholesterol, total and direct bilirubin, uric acid, total protein and albumin levels.
Number of subjects with abnormal Urinalysis parameters as a measure of safety assessed by dipstick test. | Up to Day 19.
  Urine sample will be collected at screening, Day 1, Day 6 and Day 19 to analyze specific gravity, pH, glucose, protein, blood and ketone bodies, and microscopic examination.
Body temperature assessment as a safety measure. | Day 0 to Day 13.
  Body temperature will be measured at screening, Day 0, Day 4 and Day 13 and sometimes when clinically indicated.
Blood pressure assessment as a safety measure. | Day 1 to Day 19.
  Clinostatic hypertension (CH) will be measured which is defined as a group of patients presenting an increase in arterial blood pressure when supine and a concurrent decrease of at least 20 millimetre of mercury (mm Hg) of Systolic blood pressure (SBP) and/or at least 10 mm Hg of Diastolic blood pressure (DBP) upon standing. SBP and DBP will be measured pre-dosing and at 2, 4, 8h post-dosing on Day 1; pre-dosing and at 2, 5, 8h post-dosing on Day 6; after discharge on Day 2, 7 and 16; post dosing on the Day 3, 5, 9, 11, 14 and 19 or early withdraw from the study.
Heart rate assessment as a safety measure. | Day 1 to Day 19.
  Heart rate will be measured pre-dosing and at 2, 4, 8h post-dosing on Day 1; pre-dosing and at 2, 5, 8h post-dosing on Day 6; after discharge on Day 2, 7 and 16; post dosing on the Day 3, 5, 9, 11, 14 and 19 or early withdraw from the study.
Electrocardiogram (ECG) assessment as a measure of safety and tolerability. | Screening and Day 19.
  12-lead ECGs will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zhang F, Li Y, Hu J, Zhong J, Li H. Population Pharmacokinetics, Safety and Tolerability of Extended-Release Bupropion and Its Three Metabolites in Chinese Healthy Volunteers. Eur J Drug Metab Pharmacokinet. 2019 Jun;44(3):339-352. doi: 10.1007/s13318-018-0537-z. PMID 30520001
- See also: Results for study 114883 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114883?search=study&b'search_terms=114883'#rs